CLINICAL TRIAL: NCT06296264
Title: Ultra-portable Ultrasound vs. Standard Ultrasound to Help Place a Peripheral Catheter in Patients at Risk of Difficult Puncture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ULTRACATHLON
Record Dates: First submitted 2024-02-22; First posted 2024-03-06 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: IV Line Placement With Ultrasound
Keywords: IV line; Ultra-portable ultrasound; Standard ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard ultrasound (Other): Comparator
  Interventions: Device: Standard ultrasound
- Ultra-portable ultrasound (Experimental)
  Interventions: Device: Ultra-portable ultrasound

INTERVENTIONS:
Device: Standard ultrasound — Placement of IV line using standard ultrasound.
  Arms: Standard ultrasound
Device: Ultra-portable ultrasound — Placement of IV line using ultra-portable ultrasound.
  Arms: Ultra-portable ultrasound

SUMMARY:
The placement of an intravenous (IV) line is a common procedure when treating adult patients in critical care, in the emergency room or in the operating room. This simple and minimally invasive procedure can sometimes be made difficult depending on the patient's morphology or their clinical condition. The procedure then becomes time-consuming, anxiety-provoking, painful and its success is uncertain.

The placement of intravenous (IV) lines under ultrasound by nurses is a rapidly developing alternative in intensive care, emergencies and the operating room.

DETAILED DESCRIPTION:
The main objective is to test the hypothesis that intravenous puncture guided by an ultraportable ultrasound machine is faster than puncture guided by a conventional ultrasound machine.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged at least 18 years old
2. Patient with an A-DIVA (Adult Difficult Intravenous Access) score > 1
3. Supported by a nurse trained in all the techniques used in the protocol
4. Patient having given free, informed and oral consent -

Exclusion Criteria:

1. Patient who has already been included in the study
2. Patient whose inclusion in the study would lead to a delay in treatment
3. Adult patient protected by law
4. Pregnant woman
5. Patient not benefiting from French Social Security system -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Intravenous (IV) line placement time | Day 0
  Time in minutes between tourniquet placement and dressing application after placement.

SECONDARY OUTCOMES:
Placement of the IV line successfully obtained from the first puncture | 12 months (estimated)
  Percentage of cases where the placement of the IV line was obtained from the first puncture
Number of skin perforations | Day 0
  Number of skin perforations required to establish the IV line
Overall success rate after 3 punctures | Day 0
  Overall success rate after 3 punctures
Use an alternative solution (central catheter) | Day 0
  Need to use an alternative solution (central catheter)
Patient satisfaction with IV line placement | Day 0
  Patient satisfaction with intravenous line placement (assessed by Likert scale)
Nurse satisfaction with IV line placement | Day 0
  Nurse satisfaction with intravenous line placement (assessed by Likert scale)
Immediate complications related to intravenous access | Day 0
  Number of immediate complications related to intravenous access, including arterial puncture and/or hematoma formation
Delayed complications related to intravenous access | Day 7
  Number of delayed complications related to intravenous access, including extravasation and/or the occurrence of infectious thrombophlebitis
Date of IV line placement and removal | Day 7
  Delays between IV line placement and removal

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph Saint Luc Hospital, Lyon, Auvergne-Rhône-Alpes, France